CLINICAL TRIAL: NCT01486329
Title: VXM01 Phase I Dose Escalation Study in Patients With Locally Advanced, Inoperable and Stage IV Pancreatic Cancer to Examine Safety, Tolerability, and Immune Response to the Investigational VEGFR-2 DNA Vaccine VXM01
Brief Title: VXM01 Phase I Dose Escalation Study in Patients With Locally Advanced, Inoperable and Stage IV Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaximm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VXM01-01-DE
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Stage IV Pancreatic Cancer
Keywords: Pancreatic cancer; Cancer vaccine; Gemcitabine; Inoperable; Gemcitabine chemotherapy; Locally advanced
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VXM01 (Experimental): Investigational anti-angiogenic live cancer vaccine
  Interventions: Biological: VXM01
- Placebo (Placebo Comparator): Placebo control
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VXM01 — Live anti-angiogenic cancer vaccine drink solution, escalating dose
  Arms: VXM01
Biological: Placebo — Drink solution
  Arms: Placebo

SUMMARY:
First-in-human phase I dose escalation study in patients with locally advanced, inoperable and stage IV pancreatic cancer to examine safety, tolerability, and immune response to the investigational VEGFR-2 DNA vaccine VXM01 to examine safety and tolerability, clinical and immunogenic response to the investigational vascular endothelial growth factor receptor 2 (VEGFR-2) DNA vaccine VXM01, and to define the maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, signed and dated
* Locally advanced, inoperable and stage IV pancreatic cancer patients according to UICC based on diagnostic imaging using computer-tomography (CT) or histological examinations
* Male or post-menopausal female
* Age above or equal to 18 years
* Chemotherapy naïve within 60 days before screening visit except gemcitabine treatment
* Karnovsky index >70
* Life expectancy >3 months
* Adequate renal, hepatic, and bone marrow function
* Absolute neutrophil count >1500/µL
* Hemoglobin >10 g/dL
* Platelets >75000/µL
* Prothrombin time and international normalized ratio (INR) <1.5 times upper limit of normal (ULN) (except under anticoagulant treatment)
* Aspartate aminotransferase <4 times ULN
* Alanine aminotransferase <4 times ULN
* Total bilirubin <3 times ULN
* Creatinine clearance estimated according to Cockcroft-Gault >30 mL/min
* Proteinuria <1 g protein on 24 h urine collection

Exclusion Criteria:

* State after pancreas resection (complete or partial)
* Resectable disease
* Drug trial participation within 60 days before screening visit
* Other previous or current malignancy except basal or squamous cell skin cancer, in situ cervical cancer, or any other cancer from which the patient has been disease-free for <2 years
* Prior vaccination with Ty21a
* Cardiovascular disease defined as:

  * Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg)
  * Arterial thromboembolic event within 6 months before randomization including:
  * Myocardial infarction
  * Unstable angina pectoris
  * Cerebrovascular accident
  * Transient ischemic attack
* Congestive heart failure New York Heart Association grade III to IV
* Serious ventricular arrhythmia requiring medication
* Clinically significant peripheral artery disease > grade 2b according to Fontaine
* Hemoptysis within 6 months before randomization
* Esophageal varices
* Upper or lower gastrointestinal bleeding within 6 months before randomization
* Significant traumatic injury within 4 weeks before randomization
* Non-healing wound, bone fracture or any history of gastrointestinal ulcers within three years before inclusion, or positive gastroscopy within 3 months before inclusion
* Gastrointestinal fistula
* Thrombolysis therapy within 4 weeks before randomization
* Bowel obstruction within the last 30 days before screening visit
* Liver cirrhosis ≥ grade B according to Child-Pugh Score-Classification
* Presence of any acute or chronic systemic infection
* Radiotherapy within 4 weeks before randomization
* Major surgical procedures, or open biopsy within 4 weeks before randomization
* Fine needle aspiration within 7 days before randomization
* Chronic concurrent therapy within 2 weeks before and during the double-blind study period with:

  * Corticosteroids (except steroids for adrenal failure) or immunosuppressive agents
  * Antibiotics
  * Bevacizumab
  * Any epidermal growth factor receptor inhibitor
  * Chemotherapy except gemcitabine before Day 10
* Multi-drug resistant gram-negative germ
* Pregnancy
* Lactation
* Inability to comply with study and/or follow-up procedures
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the study results or render the patient at high risk for treatment complications
* Women of childbearing potential
* Any history of drug hypersensitivity
* Any condition which results in an undue risk for the patient during the study participation according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-12; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 38 days
  Number of dose-limiting toxicities and maximum tolerated dose

SECONDARY OUTCOMES:
Immune response | Up to 24 months
  Number of immune positive patients
Tumor staging | Up to 24 months
  Tumor staging according to RECIST criteria
Tumor perfusion | Up to 24 months
  Tumor perfusion determined by DCE-MRI

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schmidt, MD, Principal Investigator — University Clinics, Heidelberg
Locations (1):
- Clinic of General Surgery, Heidelberg, Germany

REFERENCES:
- [Derived] Wick W, Platten M, Wick A, Hertenstein A, Radbruch A, Bendszus M, Winkler F. Current status and future directions of anti-angiogenic therapy for gliomas. Neuro Oncol. 2016 Mar;18(3):315-28. doi: 10.1093/neuonc/nov180. Epub 2015 Oct 12. PMID 26459812
- [Derived] Niethammer AG, Lubenau H, Mikus G, Knebel P, Hohmann N, Leowardi C, Beckhove P, Akhisaroglu M, Ge Y, Springer M, Grenacher L, Buchler MW, Koch M, Weitz J, Haefeli WE, Schmitz-Winnenthal FH. Double-blind, placebo-controlled first in human study to investigate an oral vaccine aimed to elicit an immune reaction against the VEGF-Receptor 2 in patients with stage IV and locally advanced pancreatic cancer. BMC Cancer. 2012 Aug 20;12:361. doi: 10.1186/1471-2407-12-361. PMID 22906006